CLINICAL TRIAL: NCT00095251
Title: A Randomized, Double-blind Trial in Ventilated ICU Patients Comparing Treatment With an Alpha2 Agonist Versus a Gamma Aminobutyric Acid (GABA)-Agonist to Determine Delirium Rates, Efficacy of Sedation, Analgesia and Discharge Cognitive Status
Brief Title: MENDS Study: Trial in Ventilated ICU Patients Comparing an Alpha2 Agonist Versus a Gamma Aminobutyric Acid (GABA)-Agonist to Determine Delirium Rates, Efficacy of Sedation, Analgesia and Discharge Cognitive Status
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Wes Ely, Professor of Medicine, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB#031089
Record Dates: First submitted 2004-11-01; First posted 2004-11-02 (Estimated); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Delirium
Keywords: Delirium; Hypnotics and Sedatives; Adrenergic alpha-Agonists; efficacy of sedation; cognitive impairment
MeSH Terms: conditions — Delirium; Cognitive Dysfunction | interventions — Dexmedetomidine; Lorazepam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexmedetomidine group (Active Comparator): Patients in the dexmedetomidine arm will receive a bolus dose of 1 μg/kg infused over 10 minutes followed by an infusion started at 0.15- 0.45 μg/kg/hr. The patient's managing physician will have the option of beginning the dexmedetomidine infusion without a bolus in circumstances where the patient's sedation level is adequate at enrollment or in the presence of baseline bradycardia /hypotension. Dexmedetomidine will be titrated every 10 minutes to achieve set target RASS score. The maximum dexmedetomidine infusion will be 1.5 μg/kg/hr.
  Interventions: Drug: Dexmedetomidine
- Lorazepam group (Active Comparator): Patients in the lorazepam arm will receive a bolus dose of 1-3 mg followed by an infusion started at 1-3 mg/hr. Lorazepam infusion will be titrated every 10 minutes to achieve set target RASS score. The maximum lorazepam infusion will be 10 mg /hr.
  Interventions: Drug: Lorazepam

INTERVENTIONS:
Drug: Dexmedetomidine — a bolus dose of 1 μg/kg infused over 10 minutes followed by an infusion started at 0.15- 0.45 μg/kg/hr. Dexmedetomidine will be titrated every 10 minutes to achieve set target RASS score. The maximum dexmedetomidine infusion will be 1.5 μg/kg/hr.
  Arms: Dexmedetomidine group
Drug: Lorazepam — Patients in the lorazepam arm will receive a bolus dose of 1-3 mg followed by an infusion started at 1-3 mg/hr. Lorazepam infusion will be titrated every 10 minutes to achieve set target RASS score. The maximum lorazepam infusion will be 10 mg /hr.
  Arms: Lorazepam group

SUMMARY:
Delirium has recently been shown as a predictor of death, increased cost, and longer length of stay in ventilated patients. Sedative and analgesic medications relieve anxiety and pain, but may contribute to patients' transitioning into delirium. It is possible that modifying the paradigm for sedation using novel therapies targeted at different receptors, such as dexmedetomidine targeting alpha2 receptors and sparing the GABA receptors, could provide efficacious sedation yet reduce the development, duration, and severity of acute brain dysfunction (delirium).

DETAILED DESCRIPTION:
Delirium occurs in 60-80% of ventilated Intensive Care Unit (ICU) patients and is independently associated with prolonged hospital stay, higher cost, a 3-fold increased risk of dying by six months and ongoing neuropsychological dysfunction. Hypothesis: Based on our preliminary work, we hypothesize that standard use of GABA agonist sedatives such as lorazepam and propofol may contribute to ICU delirium and its attendant untoward clinical outcomes. An alternative sedation strategy targeting alpha2 receptors and sparing GABA receptors (dexmedetomidine) might reduce delirium, provide adequate sedation, reduce analgesic requirement, and concurrently improve cognitive performance.

Long-term objective: To standardize and compare different strategies of sedation and analgesia for ventilated ICU patients in order to optimize their clinical outcomes focusing on delirium and the long-term neuropsychological dysfunction of ICU survivors.

Specific Aims:

* to study prevalence and duration of delirium in critically ill patients using differential exposure to alpha2 vs. GABA receptor agonists while evaluating efficacy of sedation and analgesia;
* to compare clinical outcomes including duration of mechanical ventilation, ICU length of stay and severity of neuropsychological dysfunction at hospital discharge; and
* to develop pharmacokinetic and pharmacodynamic models for dexmedetomidine and lorazepam when used for up to 5 days in ICU patients.

Relationship to anesthesiology: We will study whether the adverse clinical outcomes associated with ICU delirium including long-term neuropsychological dysfunction can be modified by the choice of psychoactive agents frequently used by anesthesiologists and intensivists.

Design: A blinded, randomized controlled trial of adult mechanically ventilated patients using a sedation strategy of dexmedetomidine ± fentanyl versus lorazepam ± fentanyl, with relevant outcomes and safety monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adult patients admitted to the medical and surgical ICU for critical illnesses requiring mechanical ventilation with expectation of being mechanically ventilated for greater than 24 hours

Exclusion Criteria:

* Subjects who are less than 18 years of age
* Subjects who are pregnant (a pregnancy test will be performed on all women of child bearing age)
* Inability to obtain informed consent from the patient or his/her surrogate
* Subjects in the ICU due to a lack of beds elsewhere in the hospital, triage issues, or withdrawal of care decisions rather than severity of illness
* Subjects admitted with alcohol or drug overdoses, suicide attempts, or alcohol/delirium tremens
* Subjects who are physiologically benzodiazepine dependent, and at risk for withdrawal syndromes
* Subjects with chronic pain syndromes on maintenance narcotics
* Subjects treated within the last 30 days with a drug or device that has not received regulatory approval as of study entry
* Subjects with a psychiatric history for which they are on neuroleptic treatment
* Subjects with documented moderate to severe dementia
* Subjects with anoxic brain injuries, strokes, neurotrauma, or neuromuscular disorders such as myasthenia gravis or Guillain Barre syndrome
* Medical team following patient unwilling to use the sedation regimens
* Subjects whose family and/or physician have not committed to aggressive support for 72 hours or who are likely to withdraw within 72 hours
* Subjects who are moribund and not expected to survive 24 hours
* Subjects not expected to survive hospital discharge due to preexisting uncorrectable medical condition
* Documented allergy to study medications
* Subjects who have either Child-Pugh Class B or C cirrhosis
* Subjects with active coronary artery disease at time of screening as defined by any recent evidence of ischemia, documented myocardial infarction, or coronary intervention within the past 6 months.
* Subjects with advanced heart block at time of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2004-08; Primary Completion 2007-08 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
achieving target sedation level | Patients will receive study drug for a maximum of 120 hours (5 days)
  The patients' managing team will set the "goal" or "target" as medically indicated using the RASS 37. A trained research nurse or physician blinded to patients' group assignment and medical management will perform measurement of the "actual" RASS level every 12 hours. Comparisons will be made between the actual and target RASS levels to determine the primary outcome measure, which is the accuracy of achieving the target sedation level.

SECONDARY OUTCOMES:
duration and severity of delirium | Patients will receive study drug for a maximum of 120 hours (5 days)
  Delirium will be measured using the CAM-ICU, every 12 hours, by the same research personnel performing the assessment of the patients' sedation level. Together, these instruments take on average only 1 to 2 minutes to perform. Delirium is said to be present if the patients are responsive to verbal stimulation with eye opening (i.e., RASS -3 or better) and are found to have an acute change or fluctuation in the course of their mental status, inattention, and either disorganized thinking or an altered level of consciousness.

CONTACTS AND LOCATIONS:
Overall Officials: E Wesley Ely, MD, MPH, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Background] Ely EW, Shintani A, Truman B, Speroff T, Gordon SM, Harrell FE Jr, Inouye SK, Bernard GR, Dittus RS. Delirium as a predictor of mortality in mechanically ventilated patients in the intensive care unit. JAMA. 2004 Apr 14;291(14):1753-62. doi: 10.1001/jama.291.14.1753. PMID 15082703
- [Background] Milbrandt EB, Deppen S, Harrison PL, Shintani AK, Speroff T, Stiles RA, Truman B, Bernard GR, Dittus RS, Ely EW. Costs associated with delirium in mechanically ventilated patients. Crit Care Med. 2004 Apr;32(4):955-62. doi: 10.1097/01.ccm.0000119429.16055.92. PMID 15071384
- [Background] Ely EW, Gautam S, Margolin R, Francis J, May L, Speroff T, Truman B, Dittus R, Bernard R, Inouye SK. The impact of delirium in the intensive care unit on hospital length of stay. Intensive Care Med. 2001 Dec;27(12):1892-900. doi: 10.1007/s00134-001-1132-2. Epub 2001 Nov 8. PMID 11797025
- [Background] Ely EW, Inouye SK, Bernard GR, Gordon S, Francis J, May L, Truman B, Speroff T, Gautam S, Margolin R, Hart RP, Dittus R. Delirium in mechanically ventilated patients: validity and reliability of the confusion assessment method for the intensive care unit (CAM-ICU). JAMA. 2001 Dec 5;286(21):2703-10. doi: 10.1001/jama.286.21.2703. PMID 11730446
- [Background] Inouye SK, Schlesinger MJ, Lydon TJ. Delirium: a symptom of how hospital care is failing older persons and a window to improve quality of hospital care. Am J Med. 1999 May;106(5):565-73. doi: 10.1016/s0002-9343(99)00070-4. PMID 10335730
- [Background] Inouye SK, Rushing JT, Foreman MD, Palmer RM, Pompei P. Does delirium contribute to poor hospital outcomes? A three-site epidemiologic study. J Gen Intern Med. 1998 Apr;13(4):234-42. doi: 10.1046/j.1525-1497.1998.00073.x. PMID 9565386
- [Background] Ostermann ME, Keenan SP, Seiferling RA, Sibbald WJ. Sedation in the intensive care unit: a systematic review. JAMA. 2000 Mar 15;283(11):1451-9. doi: 10.1001/jama.283.11.1451. PMID 10732935
- [Background] Marcantonio ER, Juarez G, Goldman L, Mangione CM, Ludwig LE, Lind L, Katz N, Cook EF, Orav EJ, Lee TH. The relationship of postoperative delirium with psychoactive medications. JAMA. 1994 Nov 16;272(19):1518-22. PMID 7966844
- [Background] Dubois MJ, Bergeron N, Dumont M, Dial S, Skrobik Y. Delirium in an intensive care unit: a study of risk factors. Intensive Care Med. 2001 Aug;27(8):1297-304. doi: 10.1007/s001340101017. PMID 11511942
- [Background] Maze M, Scarfini C, Cavaliere F. New agents for sedation in the intensive care unit. Crit Care Clin. 2001 Oct;17(4):881-97. doi: 10.1016/s0749-0704(05)70185-8. PMID 11762266
- [Background] National Research Council (US) Committee on Future Directions for Cognitive Research on Aging; Stern PC, Carstensen LL, editors. The Aging Mind: Opportunities in Cognitive Research. Washington (DC): National Academies Press (US); 2000. Available from http://www.ncbi.nlm.nih.gov/books/NBK44833/ PMID 20669496
- [Background] Maldonado J, Wysong A, Starre Pvd, Block T. Postoperative Sedation and the Incidence of ICU Delirium in Cardiac Surgery Patients. ASA. 2004;Abstract and Poster Presentation.
- [Derived] Stollings JL, Thompson JL, Ferrell BA, Scheinin M, Wilkinson GR, Hughes CG, Shintani AK, Ely EW, Girard TD, Pandharipande PP, Patel MB. Sedative Plasma Concentrations and Delirium Risk in Critical Illness. Ann Pharmacother. 2018 Jun;52(6):513-521. doi: 10.1177/1060028017753480. Epub 2018 Jan 24. PMID 29363356
- [Derived] Pandharipande PP, Sanders RD, Girard TD, McGrane S, Thompson JL, Shintani AK, Herr DL, Maze M, Ely EW; MENDS investigators. Effect of dexmedetomidine versus lorazepam on outcome in patients with sepsis: an a priori-designed analysis of the MENDS randomized controlled trial. Crit Care. 2010;14(2):R38. doi: 10.1186/cc8916. Epub 2010 Mar 16. PMID 20233428
- [Derived] Pandharipande PP, Pun BT, Herr DL, Maze M, Girard TD, Miller RR, Shintani AK, Thompson JL, Jackson JC, Deppen SA, Stiles RA, Dittus RS, Bernard GR, Ely EW. Effect of sedation with dexmedetomidine vs lorazepam on acute brain dysfunction in mechanically ventilated patients: the MENDS randomized controlled trial. JAMA. 2007 Dec 12;298(22):2644-53. doi: 10.1001/jama.298.22.2644. PMID 18073360
- See also: This is an educational website on delirium in the ICU. — http://www.ICUdelirium.org